CLINICAL TRIAL: NCT06629246
Title: A Randomized Controlled Trial to Evaluate the Efficacy and Safety of Pogejiuxin Decoction Combination of Conventional Treatment for Heart Failure with Preserved Ejection Fraction(HFpEF)
Brief Title: Pogejiuxin Decoction Combination of Conventional Western Medicine for the Treatment of Heart Failure with Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Traditional Chinese Medicine Hospital (Other)
Collaborators: Chongqing Science and Technology Commission (Other); Chongqing Health and Family Planning Commission (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ky-17
Record Dates: First submitted 2024-09-23; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure, Diastolic (HFpEF)
Keywords: Pogejiuxin Decoction; heart failure with preserved ejection fraction
MeSH Terms: conditions — Heart Failure; Heart Murmurs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): The control group will receive conventional heart failure treatment, which may include pharmacological therapies such as diuretics, ACE inhibitors/ARBs, beta-blockers, or aldosterone receptor antagonists, based on the clinical requirements of the condition, for a treatment period of 7 days.
  Interventions: Drug: Conventional heart failure treatment
- intervention group (Active Comparator): The intervention group will receive Pogejiuxin Decoction orally, in addition to the treatment protocol given to the control group.The specific medicinal formula is as follows: Processed Aconite 60g (decocted initially for 1 hour), Dried Ginger 60g, Honey-fried Licorice 60g, Cornus officinalis 60g, Ginseng 30g (decocted separately), Raw Dragon Bone 30g (decocted initially for 1 hour), Raw Oyster Shell 30g (decocted initially for 1 hour), Living Magnetite 30g, for a total of 7 prescriptions. Usage: Uniformly decocted with a herbal medicine decoction machine to obtain the medicinal liquid, one prescription per day, taken twice daily in the morning and evening, each time 100ml, for a continuous treatment of 7 days.
  Interventions: Drug: Pogejiuxin decoction combined with conventional heart failure treatment

INTERVENTIONS:
Drug: Conventional heart failure treatment — Conventional heart failure treatment, which may include pharmacological therapies such as diuretics, ACE inhibitors/ARBs, beta-blockers, or aldosterone receptor antagonists, based on the clinical requirements of the condition.
  Arms: control group
Drug: Pogejiuxin decoction combined with conventional heart failure treatment — In addition to receiving standard heart failure treatment, patients are also administered Pogejiuxin Decoction.The formula of Pogejiuxin Decoction is as follows : Processed Aconite 60g (decocted initially for 1 hour), Dried Ginger 60g, Honey-fried Licorice 60g, Cornus officinalis 60g, Ginseng 30g (decocted separately), Raw Dragon Bone 30g (decocted initially for 1 hour), Raw Oyster Shell 30g (decocted initially for 1 hour), Living Magnetite 30g, for a total of 7 prescriptions. Usage: Uniformly decocted with a herbal medicine decoction machine to obtain the medicinal liquid, one prescription per day, taken twice daily in the morning and evening, each time 100ml, for a continuous treatment of 7 days.
  Arms: intervention group

SUMMARY:
The objective of this study is to investigate the potential of Pogejiuxin Decoction to enhance the efficacy and mitigate the adverse effects associated with conventional treatment in patients with heart failure and preserved ejection fraction(HFpEF), thereby establishing a foundation for its clinical application in managing HFpEF.

DETAILED DESCRIPTION:
This study recruits patients with heart failure and preserved ejection fraction(HFpEF), randomly assigning them to either the intervention group or the control group. The control group will receive the standard heart failure treatment protocol, while the intervention group will take Pogejiuxin Decoction orally in addition to the control group's treatment. The study will compare the degree of symptom improvement, relevant auxiliary examination indicators, traditional Chinese medicine syndrome scores, and adverse reaction differences between the two groups, providing a clinical basis for the further enhancement of HFpEF treatment with the combination of Pogejiuxin Decoction and conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients with heart failure who meet the diagnostic criteria of China Guidelines for the Diagnosis and Treatment of Heart Failure 2018 and have grade II-IV heart function;
2. Inpatients who meet the diagnostic criteria for heart failure in TCM Internal Medicine(2012 edition);
3. Patients who meet the diagnostic criteria for HfpEF by heart color ultrasound;
4. Patients who sign informed consent and take the test voluntarily.

Exclusion Criteria:

1. Patients who do not meet the inclusion criteria.
2. Patients with severe hepatic or renal impairment (ALT/AST > 3 times the upper limit or serum creatinine levels > 265 umol/L or serum potassium > 5.5 mmol/L).
3. Patients with severe cerebrovascular, hematological, neurological diseases, or malignant tumors that require special treatment during the study period and may affect the judgment of heart failure treatment efficacy.
4. Patients with severe pneumonia, serious infections, or acute exacerbation of chronic obstructive pulmonary disease.
5. Pregnant or nursing women.
6. Patients with psychiatric abnormalities or unwilling to cooperate.
7. Patients allergic to the components of Pogejiuxin Decoction.
8. Patients undergoing coronary intervention, cardiac pacemaker implantation, placement of cardiac assist devices, or other treatments during the trial period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | From enrollment to the end of treatment at 7 days
  NT-proBNP, secreted by cardiac muscle cells, serves as a biomarker that reflects cardiac function. Under normal conditions, the body contains a small amount of NT-proBNP. However, in cases of heart failure, the levels of NT-proBNP increase, making it one of the indicators for diagnosing heart failure and assessing the effectiveness of heart failure treatment. The specific diagnostic criteria are as follows:
  For patients under 50 years of age: over 450 ng/L; For patients aged from 50 to 75: over 900 ng/L; For patients over 75 years of age: over 1800 ng/L; For patients with impaired renal function (glomerular filtration rate over 60 mL/min): over 1200 ng/L.
Echocardiography(LVEF, LVEDD and LVESD) | From enrollment to the end of treatment at 7 days
  Echocardiography is used to assess cardiac function. LVEF Left ventricular ejection fraction (LVEF) is the most commonly used indicator to evaluate left ventricular systolic function in clinical practice. LVEF is calculated from the measurements of end-diastolic volume (EDV) and end-systolic volume (ESV), using the following formula:LVEF = (EDV - ESV) / EDV × 100%. An LVEF of less than 52% in males and less than 53% in females suggests abnormal left ventricular systolic function. An LVEF between 40% and 52% indicates mildly reduced left ventricular systolic function, 30% to 40% indicates moderately reduced function, and less than 30% indicates severely reduced function.
  LVEDD and LVESD In males, a left ventricular end-diastolic diameter (LVEDD) over 55 mm and in females over 50 mm, and a left ventricular end-systolic diameter (LVESD) over 37 mm in males and over 35 mm in females, suggest left ventricular dilation and impaired left ventricular function.
hs-CRP | From enrollment to the end of treatment at 7 days
  High-sensitivity C-reactive protein (hs-CRP) is one of the most potent predictors of cardiovascular risk events, with the following clinical implications:
  A level of under 1 mg/L indicates low risk; A level of 1-3 mg/L indicates moderate risk; A level above 3 mg/L indicates high risk.
Inflammatory Factors(TNF-α, IL-6, and IL-8) | From enrollment to the end of treatment at 7 days
  Clinical practice has confirmed that levels of inflammatory cytokines such as TNF-α, IL-6, and IL-8 are elevated in patients with heart failure compared to the general population. These inflammatory factors can further exacerbate myocardial damage and participate in the process of ventricular remodeling. Therefore, monitoring TNF-α, IL-6, and IL-8 can be used to assess the condition of patients with heart failure. Elevated levels of TNF-α over 5 ng/L (bioactivity assay), IL-6 over 10 ng/L, and IL-8 over 21.3 μg/L (ELISA method) suggest the presence of inflammation in the body.
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | From enrollment to the end of treatment at 7 days
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a widely used instrument for assessing health-related quality of life in patients with heart failure (HF). It evaluates quality life of patients across three domains: physical, emotional, and other. The questionnaire consists of 21 items, with responses rated on a scale from zero to five, indicating none (0 points), very little (1 point), a little (2 points), moderate (3 points), quite a bit (4 points), and severe (5 points). The scores of all items are summed up, with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
Traditional Chinese Medicine (TCM) Symptom Score | From enrollment to the end of treatment at 7 days
  According to the Guiding Principles for Clinical Research of New Drugs in Traditional Chinese Medicine. The Traditional Chinese Medicine (TCM) symptoms are categorized into primary and secondary symptoms and are scored based on their severity. Primary symptoms include palpitations, fatigue, dyspnea, and lower limb edema, each rated on a scale of four levels: none (0 points), mild (2 points), moderate (4 points), and severe (6 points). Secondary symptoms include lethargy, abdominal distension, oliguria, spontaneous sweating, and dull complexion/cyanosis of lips and nails, each rated on a scale of four levels: none (0 points), mild (1 point), moderate (2 points), and severe (3 points). The total score from all items represents the TCM symptom score.The higher the score, the more severe the symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Liu L, Mo Y, Wu B, Yu Z, Sun B. Effect of Traditional Chinese Medicine Poge Heart-Saving Decoction on Cardiac Function in Heart Failure Rat Model. Evid Based Complement Alternat Med. 2020 Dec 3;2020:8762509. doi: 10.1155/2020/8762509. eCollection 2020. PMID 33628294
- [Background] Li X, Zhang J, Huang J, Ma A, Yang J, Li W, Wu Z, Yao C, Zhang Y, Yao W, Zhang B, Gao R; Efficacy and Safety of Qili Qiangxin Capsules for Chronic Heart Failure Study Group. A multicenter, randomized, double-blind, parallel-group, placebo-controlled study of the effects of qili qiangxin capsules in patients with chronic heart failure. J Am Coll Cardiol. 2013 Sep 17;62(12):1065-1072. doi: 10.1016/j.jacc.2013.05.035. Epub 2013 Jun 7. PMID 23747768
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794